CLINICAL TRIAL: NCT03531450
Title: Central and Peripheral Effects of Cognitive Behavioral Therapy on Brain-Gut Axis Signaling in Gastroparetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Braden Kuo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Partners Protocol ID Pending
Record Dates: First submitted 2018-04-25; First posted 2018-05-21 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Gastroparesis
Keywords: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): Patients in the cognitive behavioral therapy group will be asked to undergo a 8-week CBT trial. An online videoconferencing link will be used to deliver CBT virtual sessions that will be approximately 60 minutes in length. Each session will be conducted by a clinical psychology doctoral student, supervised by a licensed psychologist. Patients will also undergo careful phenotyping pre- and post intervention with brain MRI, AFT, and NDT.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Treatment sessions will use active, structured techniques to alter distorted thoughts, with a focus on acquiring and practicing cognitive and emotional modulatory skills. In particular, cognitive restructuring is used to help patients recognize the relationships between thoughts, feelings, and behaviors. Patients learn to identify, evaluate, and challenge negative thoughts. Patients will also learn behavioral strategies to decrease avoidance behavior and increase toleration of physical sensations.

SUMMARY:
This is a single-center pilot study to be conducted at Massachusetts General Hospital. The purpose of this study is to examine the non-pharmacological impact of Cognitive Behavioral Therapy (CBT) on gastroparesis symptoms and other clinical co-comorbidities such as pain, depression, anxiety, and catastrophizing. CBT trial patients will undergo careful phenotyping pre- and post- intervention with brain MRI, autonomic function test (AFT), gastric emptying scintigraphy (GES), and nutrient drink test (NDT) to determine the impact of CBT on these metrics in patients with gastroparesis. Characterization of these relationships or lack thereof can help guide future development of more targeted approaches and optimize treatment strategies for gastroparesis.

DETAILED DESCRIPTION:
This randomized, controlled trial will examine the effects of cognitive behavioral therapy (CBT) on gastroparesis symptoms (including pain related brain circuitry). CBT reduces pain intensity, negative affect, and disability among patients with chronic pain, though there is a good deal of individual variability in treatment effects. Treatment gains following CBT are maintained or enhanced at 6 to 12-month follow-up. This study will examine the brain circuitry underlying these effects. In addition, as measures of gastroparesis symptoms and pain are correlated with other, more general, measures of negative affect (e.g., depression, anxiety), we will evaluate the specificity of the hypothesized effects by running the proposed statistical models both with and without inclusion of these conceptually overlapping factors. Based on pervious findings and published data, we expect that treatment-associated changes in pain and depression will likely share 10-20% of their variance.

Treatment sessions will use active, structured techniques to alter distorted thoughts, with a focus on acquiring and practicing cognitive and emotional modulatory skills. CBT is based on a pain self-management paradigm, and involves the identification and reduction of maladaptive pain-related cognitions (i.e., catastrophizing) using techniques such as relaxation, thought-stopping, distraction, etc. CBT prominently emphasizes in-vivo practice during each session, and features home practice using written exercises. In particular, cognitive restructuring is used to help patients recognize the relationships between thoughts, feelings and behaviors. Patients learn to identify, evaluate, and challenge negative thoughts. In our protocol, each of the 8 weekly sessions will last for approximately 90 minutes and will be conducted or supervised by a trained psychologist. Following CBT, negative emotions are no longer closely linked to pain, suggesting that CBT provides patients with the skills to modulate and buffer their negative emotions such as catastrophizing.

Subjects will undergo pre- and post-treatment testing through a variety of methods including brain MRI with associated physiological data, autonomic function test (AFT), gastric emptying scintigraphy (GES), and nutrient drink test (NDT) to determine the impact of CBT on these metrics in patients with gastroparesis. Characterization of these relationships or lack thereof can help guide future development of more targeted approaches and optimize treatment strategies for gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 - 65 years old (inclusive)
2. Symptoms of gastroparesis of at least 12 weeks duration (do not have to be continuous) with varying degrees of nausea, vomiting, early satiety, and/or post-prandial fullness
3. An idiopathic etiology
4. GES of solids using 4 hours Egg Beaters® protocol within the last 2 years with either:

   - Abnormal gastric emptying rate defined as an abnormal 2 hour (>60% retention) and/or 4 hour (>10% retention) result based on a 4 hour scintigraphic low fat Egg Beaters® gastric emptying study.
5. Body mass index (BMI) ≥ 17.5 kg/m2
6. Have not previously received CBT for coping with chronic illness
7. Have access to a computer with internet access
8. Speak, write, and understand English
9. On stable doses of any medication for 30 days prior to entering the study (exceptions are psychotropic, opioids, and/or illicit drugs) and agrees not to change medications or dosages during the study period.

Exclusion Criteria:

1. Inability to comply with or complete GES test (including allergy to eggs)
2. Use of narcotic analgesics greater than three days per week
3. Presence of other conditions that could explain the patient's symptoms:

   * Pyloric or intestinal obstruction as determined by endoscopy, upper GI series or abdominal CT scan
   * Active inflammatory bowel disease
   * Known eosinophilic gastroenteritis or eosinophilic esophagitis
   * Primary neurological conditions that could cause nausea and/or vomiting such as increased intracranial pressure, space occupying or inflammatory/infectious lesions
   * Acute liver failure
   * Acute renal failure
   * Chronic renal failure (serum creatinine >3 mg/dL) and/or on hemodialysis or peritoneal dialysis
   * Prior gastric surgery to restore function or relieve GI symptoms including total or subtotal (near complete) gastric resection, esophagectomy, gastrojejunostomy, or gastric bypass, gastric sleeve, pyloroplasty, pyloromyotomy. Note: patients with prior (Nissen, Dor, or Toupet) fundoplication will be eligible for enrollment.
   * Subject has current evidence of duodenal ulcer, gastric ulcer, diverticulitis, active GERD or infectious gastroenteritis.
   * Any acute gastrointestinal process.
   * Any other plausible structural or metabolic cause
   * Any condition, which in the opinion of the investigator, would interfere with study requirements
4. Inability to provide informed consent
5. BMI more than 32 and/or weight > 235 lbs. (limits of the MRI table)
6. Enteral or parenteral feeding
7. Epilepsy or a prior history of seizures
8. Pregnancy or nursing
9. Psychotherapy initiated in the last 8 weeks
10. Contraindications for MRI: High magnetic fields may pose a serious health hazard to subjects with implanted ferromagnetic objects. Every subject in this study will be carefully screened before entering the high magnetic field shielded room to collect a precise outline of the subject's medical history. Subjects with the following characteristics/disease will not be eligible to participate in the study:

    * History of Head Trauma
    * Any metallic implants (e.g. braces or permanent retainers)
    * Tattoos with metallic ink above the nipple line
    * Surgical Aneurysm Clips
    * Cardiac Pacemaker
    * Prosthetic Heart Valve
    * Neurostimulator
    * Implanted pumps
    * Cochlear Implants
    * Metal rods, Plates
    * Screws
    * Recent Previous Surgery
    * IUD
    * Hearing Aid
    * Dentures (which might create NMR artifacts)
    * Metal Injury to eyes
    * Pregnancy or plans to become pregnant
    * Breast Feeding
    * Meniere's Disease
    * Transdermal (skin) patches such as NicoDerm (nicotine for tobacco dependence), Transderm Scop, or Ortho Evra (birth control)
    * Claustrophobia
    * Suicidal ideation as indicated from the HADS

All concomitant medications taken during the study will be recorded in the case report form, along with dosage information and start and stop dates. Patients requiring excluded drugs will be discontinued from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Patient Assessment of Upper Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) | Up to 12 weeks
  One of the primary endpoints will be change in gastroparesis symptom severity by the Gastroparesis Cardinal Symptom Inventory (GCSI). The GCSI is comprised of three subscales: post-prandial fullness/early satiety, nausea/vomiting, and bloating. A one-point decrease in the GCSI has been validated to indicate clinically significant improvement.

SECONDARY OUTCOMES:
Gastrointestinal symptom assessment via Short Form 36 Health Survey | Up to 12 weeks
Gastrointestinal symptom assessment via Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life | Up to 12 weeks
  Another primary endpoint will be a change in gastroparesis-related quality of life, as assessed by the Patient Assessment of Gastrointestinal Symptoms - Quality of Life (PAGI-QOL).
Gastrointestinal symptom assessment via Rome III Diagnostic Questionnaire for Adult Functional GI Disorders | Up to 12 weeks
Gastrointestinal symptom assessment via Hospital Anxiety and Depression Scale | Up to 12 weeks
  The HADS contains subscales for anxiety and depression (7 items each, scored 0-3) and will be used to explored as a potential moderator of treatment outcome.
Gastrointestinal symptom assessment via Patient Health Questionnaire | Up to 12 weeks
Gastrointestinal symptom assessment via PainDETECT | Up to 12 weeks
  The questionnaire is scored on a scale of 0-38. Scores of 0-12 indicate that a neuropathic pain component is unlikely (>15%), scores of 13-18 are ambiguous, however a neuropathic pain component can be present, and scores of 18-36 indicate that a neuropathic pain component is likely (>90%). We will use the PainDETECT to explore neuropathic pain severity as a potential moderator of treatment outcome
Gastrointestinal symptom assessment via Pain Catastrophizing Scale | Up to 12 weeks
  This questionnaire assesses a patient's level of pain-related worry across three areas: rumination, helplessness, and magnification. The questionnaire lists 12 reactions to pain and asks subjects to identify how often they have these reactions on a scale of 0-4, for a maximum possible total score of 56. We will use the Pain Catastrophizing Scale to explore pain-related worry as a potential mechanism of change in CBT.
Gastrointestinal symptom assessment via Neuropathy Total Symptoms Score | Up to 12 weeks
Gastrointestinal symptom assessment via PTSD Questionnaire - PCL-5 | Up to 12 weeks
Gastrointestinal symptom assessment via Brief Pain Inventory | Up to 12 weeks
  This questionnaire assesses pain in gastroparesis patients
Gastrointestinal symptom assessment via Early Life Trauma Inventory Self Report - Short Form | Up to 12 weeks
Gastrointestinal symptom assessment via Coping Strategies Questionnaire | Up to 12 weeks
  This questionnaire assess an array of pain coping methods such as distraction
Gastrointestinal symptom assessment via Pain Self-Efficacy Questionnaire | Up to 12 weeks
  This questionnaire measures perceived self-efficacy for managing various aspects of pain.
Gastrointestinal symptom assessment via Eysenck Personality Inventory | Up to 12 weeks
Gastrointestinal symptom assessment via Perceived Stress Scale | Up to 12 weeks
Structural fMRI, resting fMRI, fMRI during catastrophizing test | Baseline, and up to 2 hours post-intervention
Multivoxel 3D Proton Resonance Spectroscopy | Baseline, and up to 2 hours post-intervention
Autonomic Function Testing (AFT) | Baseline, and up to 1 hour post-intervention
  We will use an autonomic functioning test (AFT) using the ANX 3,0 autonomic monitoring system. Autonomic parameters computed by the ANX 3.0 system included the following parameters: sympathetic activity (LFa), parasympathetic activity (RFa), and sympathovagal balance (LFa/RFa). We will use the AFT to explore autonomic function as a potential mechanism of change in CBT.
Abdominal Quantitative Sensory Testing (QST) | Baseline, and up to 1 hour post-intervention
  The QST assesses subject response to sharp prick and pressure sensations on the arm, finger, and abdomen. We will examine temporal summation from the abdominal QST as a potential mechanism of change in CBT.
Electrogastrogram acquired during MRI scans | Baseline, and up to 2 hour post-intervention
Electrocardiogram acquired during MRI scans | Baseline, and up to 2 hour post-intervention
Respiration during MRI scans | Baseline, and up to 2 hour post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Braden Kuo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States